CLINICAL TRIAL: NCT07274423
Title: Clinical Value of Deep Learning Reconstruction Technology in Ankle MRI
Status: Recruiting | Type: Observational
Sponsor: Lian Yang (Other)
Responsible Party: Sponsor-Investigator, Lian Yang, Director, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Other Study IDs: 2025-0802
Record Dates: First submitted 2025-11-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Ankle Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- scanning using AI-based ankle MRI sequences
- scanned using non-AI ankle MRI sequences

SUMMARY:
By enrolling patients who underwent ankle MR(Magnetic Resonance) examinations at our center and using randomized allocation, the patients were divided into a study group and a control group. The study group underwent scanning using AI-based(Artificial Intelligence-based) ankle MRI sequences, while the control group was scanned using non-AI ankle MRI sequences.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing ankle MRI at Wuhan Union Hospital from August 2025 to August 2026;
2. Aged > 18 years old;
3. Patients who agree to participate in the study and provide signed informed consent;
4. Presence of a clear history of ankle trauma and related symptoms requiring MRI for diagnosis or evaluation.

Exclusion Criteria:

1 .Patients with MR examination contraindications (e.g., implanted metal devices or severe claustrophobia); 2. Patients with prior ankle surgery; 3. Patients who failed to complete MR examination or whose image quality was insufficient for diagnostic purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a clear history of ankle trauma
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | immediately after procedure
  Patient satisfaction will be evaluated using a Likert scale with the following scoring criteria:5 - Very Satisfied;4 - Satisfied;3 - Neutral;2 - Dissatisfied;1 - Very Dissatisfied.

SECONDARY OUTCOMES:
objective image measurements (signal-to-noise ratio) | one week
total scan time | During procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital，Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei, China